CLINICAL TRIAL: NCT04933539
Title: A Phase 2 Adaptive Study of Subcutaneous Daratumumab, Once Weekly Carfilzomib, and Dexamethasone (DKd) in Patients With High-Risk Smoldering Multiple Myeloma
Brief Title: Subcutaneous Daratumumab, Once Weekly Carfilzomib, and Dexamethasone (DKd) in Patients With High-Risk Smoldering Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210024; 21-C-0024
Record Dates: First submitted 2021-06-18; First posted 2021-06-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Multiple Myeloma
Keywords: anti-CD38 monoclonal antibody; Proteasome Inhibitor; Anti-Myeloma Activity; Immunomodulatory Agents; Combination Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; carfilzomib; daratumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Daratumumab SC (Cycles 1-2: Days 1, 8, 15, 22; Cycles 3-6: Days 1, 15; Cycles =7: Days 1 of the 28-day cycle); Carfilzomib IV (Days 1, 8, 15 of the 28-day cycle); Dexamethasone PO/IV (Days 1, 8, 15, 22 of the 28-day cycle)
  Interventions: Drug: Dexamethasone; Drug: Carfilzomib; Biological: Daratumumab

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone PO/IV (for Cycles 1-4: Dexamethasone 40 mg IV/PO on days 1, 8, 15, 22; for Cycles =5: Dexamethasone 20 mg IV/PO on days 1, 8, 15, 22); for up to 12 cycles
Drug: Carfilzomib — Carfilzomib IV (for Cycles 1-2: 20 mg/m2 IV on day 1, 56 mg/m2 IV on days 8, 15; Cycles =2: 56/m2 IV on days 1, 8, 15); for up to 12 cycles
Biological: Daratumumab — Daratumumab SC 1800 mg (Cycles 1-2: Days 1, 8, 15, 22; Cycles 3-6: Days 1, 15; Cycles =7: Days 1 of the 28-day cycle); up to 36 cycles total

SUMMARY:
Background:

Multiple myeloma (MM) is a tumor in which malignant plasma cells accumulate in the bone marrow. It can cause organ damage and is not curable. Researchers want to see if a combination drug treatment can help.

Objective:

To try to prevent or slow down developing MM and its associated organ damage by treating it while still in the smoldering phase with a mix of drugs known as DKd.

Eligibility:

People ages 18 and older with smoldering MM that is at high risk of converting to symptomatic MM.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Bone survey (x-rays of their bones)

Spinal magnetic resonance imaging

Bone marrow biopsy (a needle is used to remove bone marrow from their hipbone)

Electrocardiogram (to check heart function)

Lung function tests

Treatment will be given in 28-day cycles. Participants will get daratumumab by injection under the skin. They will get carfilzomib intravenously (IV) through a tube inserted in a vein. They will get dexamethasone as oral tablets or as an IV. They will get all 3 drugs for 8 or 12 cycles. Then they will get daratumumab alone for up to 24 cycles. They may have stem cells collected.

Participants will have frequent study visits. At these visits, they will repeat some screening tests. They will complete questionnaires. They will have imaging scans. For these scans, they may receive an oral or IV contrast.

Participants will have a follow-up visit 30 days after treatment ends. Then they will have visits every 3-12 months. They will be followed on this study for life.

DETAILED DESCRIPTION:
Background:

Smoldering multiple myeloma (SMM) is a precursor condition to MM defined by the clinical parameters of M-protein >=3.0 g/dL or bone marrow plasma cells >=10%, and absence of end organ disease.

Patients with high-risk SMM have a risk of progression to MM of 72-75% in 5 years with median time to progression of <2 years.

The current standard of care for SMM is close follow-up without treatment, until symptomatic MM develops. However, International Myeloma Working Group (IMWG) recommends Preventive clinical trials need to be considered for patients with high risk smoldering myeloma.

Carfilzomib is a proteasome inhibitor and daratumumab is an anti-CD38 monoclonal antibody, both with potent anti-MM effects.

Objectives:

To assess the remission rate of daratumumab, carfilzomib, and dexamethasone (DKd) in patients with high-risk (HR) smoldering multiple myeloma (SMM) by determining the minimal residual disease (MRD) negative complete response (CR) rate by up to 12 cycles of induction therapy using flow cytometry.

Eligibility:

SMM according to the IMWG definition; i.e.:

Serum M-protein >=3 g/dl and/or bone marrow plasma cells >=10 % and <60%

Absence of anemia: Hemoglobin >10 g/dl

Absence of renal failure: serum creatinine <2.0 mg/dL.

Absence of hypercalcemia: Ca <10.5 mg/dl or 2.62 mmol/L

Absence of lytic bone lesions

<=1 focal lesion on MRI

Involved/un-involved light chain ratio <100

High-risk SMM per Mayo Clinic, Spanish PETHEMA, or the Rajkumar, Landgren, Mateos criteria

Age >=18 years

Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Adequate laboratory parameters

Design:

Single arm trial of combination therapy (daratumumab, carfilzomib, and dexamethasone) followed by daratumumab maintenance monotherapy (DKd-D) for high-risk SMM.

Participants will receive 8 cycles of DKd induction combination therapy. After 8 cycles, participants who have not attained an MRD negative remission will receive 4 additional cycles of DKd. Each cycle consists of 28-days.

After 4 cycles of induction therapy, transplant eligible participants may choose to undergo stem cell collection for storage.

After induction with DKd, participants will receive daratumumab maintenance therapy for 24 cycles.

Participants will have routine blood work with SPEP and free light chains at the start of each cycle during the induction phase. Laboratory evaluations may be spread out to every 3-6 months during the maintenance and follow-up phases.

Pre-treatment, post-treatment and follow-up bone marrow biopsies will be obtained for confirmation of diagnosis, response and correlative studies.

Participants will also undergo evaluation for MRD at regular interval time points, using multi-parametric flow cytometry, FDG PET-CT, and Diffusion Weighted Whole Body (DW-MRI).

The statistical analysis of the primary endpoint, MRD negativity, will be performed at the end of induction therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed smoldering multiple myeloma (SMM) based on the International Myeloma Working Group Criteria:

  * Serum M-protein >=3 g/dl and/or bone marrow plasma cells >=10 % and <60%
  * Absence of anemia: hemoglobin >10 g/dl
  * Absence of renal failure: serum creatinine <2.0 mg/dL
  * Absence of hypercalcemia: Ca <10.5 mg/dl or 2.62 mmol/L
  * Absence of lytic bone lesion on X-ray, CT, or PET/CT and not more than 1 lesion on spinal MRI (NOTE: At the discretion of the investigator, PET/CT may replace MRI in patients who have a contraindication to MRI.)
  * Involved/un-involved light chain ratio must be < 100 (unless involved light chain is <=10 mg/dL)
* Measurable disease within the past 4 weeks defined by any one of the following:

  * Serum monoclonal protein >= 0.5 g/dl
  * Urine monoclonal protein >200 mg/24 hour
  * Serum immunoglobulin free light chain >10 mg/dL AND abnormal kappa/lambda serum free light chain ratio (reference 0.26-1.65)
  * Because the primary endpoint is MRD (-) remission rate, per the discretion of the Principal Investigator, patients without measurable disease in the serum (e.g., Mspike <0.5 g/dL) may also be enrolled. This is in line with the most recent IMWG MM response criteria.
* Age >=18 years.
* ECOG performance status <=2
* Patients must have adequate organ and marrow function as defined below:

  * absolute neutrophil count (ANC) >=1.0 K/uL

NOTE: At the discretion of the investigator, patients with an ANC of 0.5 K/uL -1.0 K/uL may also be enrolled if clinically appropriate (e.g., patients with a baseline neutropenia that is chronic and that does not cause complications).

* platelets >=75 K/uL
* hemoglobin > =8 g/dL, for anemia not due to MM (transfusions are permissible)
* total bilirubin = <1.5 X institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) =<3.0 X institutional upper limit of normal
* creatinine within normal institutional limits, OR
* If creatinine is outside of the normal limits, then creatinine Clearance (CrCl) or Egfr (estimated glomerular filtration Rate) >=40 ml/min calculated by Cockcroft-Gault method, modification of diet in renal disease (MDRD), or the chronic kidney disease (CKD)-epidemiology collaboration (EPI) (institutional standard) equations.

  -In addition to having SMM, patients must also be classified as high-risk SMM per at least one of three criteria below:
* Criteria 1: Mayo Clinic 2018, high-risk defined with two of the following:

  * Bone marrow plasmacytosis >=20%,
  * Serum monoclonal protein >=2 g/dL
  * Serum free light chain ratio of >=20
* Criteria 2: Spanish PETHEMA, high-risk defined as:
* Immunoparesis (depression of one of the uninvolved immunoglobulin isotypes in the total serum immunoglobulin assay, AND

  -->=95% aberrant plasma cells on bone marrow aspirate flow cytometry
* Criteria 3: Rajkumar, Landgren, Mateos may also be used to define high risk disease, namely clonal bone marrow plasma cells >=10% AND any one or more of the following:

  * Serum M protein >=30g/L,
  * IgA SMM,
  * Immunoparesis with reduction of 2 uninvolved immunoglobulin isotypes,
  * Serum involved/uninvolved FLC ratio >=8 (but <100),
  * Progressive increase in M protein level (evolving type of SMM; increase in serum M protein by >=25% on 2 successive evaluations within a 6-month period),
  * Clonal BMPCs 50%-60%,
  * Abnormal PC immunophenotype ( (Bullet)95% of BMPCs are clonal) and reduction of >=1 uninvolved immunoglobulin isotypes,
  * t(4;14) or del(17p) or 1q gain,
  * Increased circulating PCs,
  * MRI with diffuse abnormalities or 1 focal lesion, AND/OR PET-CT with focal lesion with increased uptake without underlying osteolytic bone destruction

    * The effects of carfilzomib and daratumumab on the developing human fetus are unknown. For this reason, individuals of child-bearing potential (IOCBP) and individuals who can father children must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 3 months after daratumumab and/or 6 months after the last dose of carfilzomib, whichever is longer. Individuals who can father children must use adequate contraception during treatment and for 3 months after stopping daratumumab and/or carfilzomib.
    * Negative serum or urine pregnancy test at screening for IOCBP.
    * Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Prior therapy for SMM. At the discretion of the investigator, exceptions might be made depending on prior treatments received and response to those treatments, provided that by the start of protocol therapy, there will be a 4-week washout period. Exceptions will not be made for patients who have received the current DKd with daratumumab maintenance regimen nor any other regimen consisting of daratumumab and a proteasome inhibitor (e.g., bortezomib, ixazomib). Treatment with corticosteroids for other indications is permitted.
* Contraindication to any concomitant medication, including support/prophylaxis for infusion reaction, antiviral, antibacterial, anticoagulation or tumor lysis given prior to therapy.
* Patient has either of the following:

  --Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal.

  ---Known moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. NOTE: Subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.
* Seropositive for human immunodeficiency virus (HIV). HIV-infected patients on effective anti-retroviral therapy with undetectable viral load for at least the 3 months prior to enrollment are eligible for this trial.
* Active hepatitis B infection. NOTE: Patients who are hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive will need to have a negative HBV PCR result before enrollment. Those with a positive PCR for hepatitis B are excluded.
* Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carfilzomib or daratumumab or other agents used in study.
* Current uncontrolled hypertension (chronic systolic blood pressures >160 mm Hg) or diabetes (chronic clinical signs/symptoms of hyperglycemia and/or an A1c value >9%).
* Significant cardiovascular disease with NYHA Class II, III or IV symptoms, or hypertrophic cardiomegaly, or restrictive cardiomegaly, or myocardial infarction within 3 months prior to enrollment, or unstable angina, or unstable arrhythmia.
* No studies of carfilzomib or daratumumab have been conducted on nursing individuals and it is not known if it is excreted in milk. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, nursing should be discontinued if the mother is treated with carfilzomib/daratumumab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, venous thromboembolic disease, hemorrhage, pulmonary fibrosis, pneumonitis, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 12 cycles
  To assess the remission rate of DKd in participants with high-risk (HR) SMM by determining the minimal residual disease (MRD) negative complete response (CR) by flow cytometry (10-5 sensitivity) rate after 12 cycles of therapy

SECONDARY OUTCOMES:
Overall Response Rate | every 6-8 weeks
  The fraction of participants who experience a PR, VGPR, CR or sCR after DKd determined by dividing the number of responders by the total evaluable patients.
Duration of Response | every 6-8 weeks
  Time from PR or better until the time of PD. Kaplan-Meier will be utilized
Biochemical and Symptomatic progression free survival (PFS) | every 6-8 weeks
  Using Kaplan-Meier method, considering those who biochemically progress or die and those who clinically progress or die, and censoring those who do not
Durability of MRD negative complete response (CR) | through 3 years post-treatment
  Sustained negative CR rate 1, 2, 3 years.
Toxicity evaluation of DKd | through 30 days post treatment
  Descriptive statistics to determine safety of receiving KRd with daratumumab maintenance
Overall survival (OS) | ongoing
  Determined using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Hill, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@All large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2021-C-0024.html